CLINICAL TRIAL: NCT03506685
Title: The Effectiveness of Dry Needling and Soft Tissue Mobilization in the Management of Pain Post Anterior Cruciate Ligament (ACL) Reconstruction: A Randomized Controlled Trial
Brief Title: Effectiveness of Dry Needling and STM on Pain Management for Anterior Cruciate Ligament Reconstruction (ACLR)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to reach agreement with PT & surgeons on protocol
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jamie Morris, principal Investigator, Keller Army Community Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 18KACH002
Record Dates: First submitted 2018-03-30; First posted 2018-04-24 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2018-04

CONDITIONS: Pain and Anterior Cruciate Ligament Reconstruction
Keywords: dry needling; ACL reconstruction; knee ROM; pain management; opioid use
MeSH Terms: conditions — Pain; Agnosia | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: 2x5 mixed model anova
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group Standard ACL protocol (No Intervention): This group will receive the standard ACL protocol rehab
- Dry needling and STM group (Experimental): This group will also receive the standard ACL protocol in addition to STM and DN
  Interventions: Other: Dry needling and STM

INTERVENTIONS:
Other: Dry needling and STM — dry needling and soft tissue mobilization
  Arms: Dry needling and STM group

SUMMARY:
The purpose of this study is to determine if dry needling (DN) and soft tissue mobilization (STM) is superior to standard treatment protocol for affecting pain, pain medication usage and measurements of range of motion (ROM) after ACL reconstruction surgery compared to a standard treatment protocol. Measurements of pain, pain medication usage, lower extremity functional scale (LEFS) and ROM will be taken day 2 post op and 1 week, 2 weeks, 3 weeks, and 4 weeks post op. It is hypothesized that the inclusion of DN and STM will acutely decrease the demand for pain medication and improve objective measurements when compared to a standard treatment protocol. Findings will potentially lead to insights as to the benefit of applying these interventions to help decrease the demand for pain medication post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 Department of Defense( DOD) beneficiaries (17 if Cadet)
* Scheduled for ACL Reconstruction Surgery

Exclusion Criteria:

* Self-Reported Pregnancy
* History of blood borne pathogens/infectious disease/active infection/metal allergy
* Bleeding disorders or currently taking anti-coagulant medications
* Participants who are not fluent in English

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Numerical pain rating scale | change from baseline, 2 days post-op, 1 week, 2 week, 3 week, 4 week
  validated outcome measure for pain ranging from 0-10

SECONDARY OUTCOMES:
Lower extremity functional scale | change from baseline, 2 days post-op, 1 week, 2 week, 3 week, 4 week
  validated measure to assess disability and function for the lower extremity on a scale of 0-80
Global rate of change | change from baseline, 2 days post-op, 1 week, 2 week, 3 week, 4 week
  validated measure of self reported overall change in injury or condition ranging from -7 to 7
knee range of motion | change from baseline, 2 days post-op, 1 week, 2 week, 3 week, 4 week
  measured with goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Keller Army Community Hospital, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
No Protected Health Information (PHI) or Personally Identifiable Information (PII) data will be share however may share outcome measures for data analysis based on subject identification.